CLINICAL TRIAL: NCT06566040
Title: Correlations Between Wheelchair Provision Time for Hospital Inpatients and Their Lengths of Stay and Costs of Hospitalization
Brief Title: Wheelchair Provision Time for Hospital Inpatients
Status: Suspended | Type: Observational
Why Stopped: Preliminary results analyzed, planning underway for next period of data collection
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: REB1030610
Record Dates: First submitted 2024-06-21; First posted 2024-08-22 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-08

CONDITIONS: Wheelchairs
MeSH Terms: interventions — Wheelchairs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wheelchair — Wheelchairs provided to hospital inpatients

SUMMARY:
In a Pilot Study, the median Wheelchair Lead Time (from when a wheelchair was ordered by an Occupational Therapist for an inpatient in the Central Zone of Nova Scotia Health to when the wheelchair arrived at the destination facility) of 119 wheelchairs was 2.98 days, with median Wheelchair Assembly Time and Wheelchair Delivery Time components of 0.98 and 1.00 days respectively. (For the over 3,000 inpatients/year for whom an order is placed, Wheelchair Delivery Time is not routinely recorded.) Reductions in Wheelchair Lead Time have the potential to speed patient mobilization (with benefits to the patient) and reduce both the patient's hospital Length of Stay and the patient-related Cost of Hospitalization. However, these potential benefits remain speculative. The objective of this project is to test the hypotheses that there are significant positive associations between Wheelchair Lead Time and both Length of Stay and the Cost of Hospitalization.

DETAILED DESCRIPTION:
The wheelchair provision process within the Central Zone of Nova Scotia Health includes the ordering, assembly, and delivery of wheelchairs from where the inventory is stored at the Nova Scotia Rehabilitation and Arthritis Centre to inpatient units at 10 sites. At discharge from hospital, the wheelchair is typically returned, cleaned and placed back in inventory. The WheelEase software that tracks components of this process was developed locally in 2001, ownership of which has transferred to the Nova Scotia Health Assistive Technology Program. The software has been periodically refined. As an indication of the volume or orders, during the 6-month period from April 1 to September 30, 2021, there were 257-277 orders per month (~13/weekday) and the WheelEase database includes over 34,000 historical wheelchair orders. People who require wheelchairs after discharge need to rent or purchase them, a process that can take several months.

During the 2022-2023 Academic Year, the Wheelchair Research Team proposed and directed a Pilot Study by a group of four final-year Industrial Engineering students. The objective of the Capstone Project was to analyze Nova Scotia Health's wheelchair provision process for inpatients in the Central Zone and provide recommendations that might improve the quality of care provided and save costs. The students used a variety of methods to collect data including regularly checking loading docks and delivery spaces, tracker sheets, Global Positioning System trackers, interviews, contextual inquiry and shadowing of wheelchair technicians, a survey of Occupational Therapists (of whom there were 64 in the Central Zone), a discrete-event simulation to compare sequencing rules for the order in which the technicians build wheelchairs and a review of the existing WheelEase database.

Among other findings from the Pilot Study, during an 11-weekday period in late January 2023, the median Wheelchair Lead Time of 119 wheelchairs was 2.98 days, with median Wheelchair Assembly Time and Wheelchair Delivery Time components of 0.98 and 1.00 days respectively. Variations among sites and the day of the week that the order was placed were identified. The average 24-hour cost of a hospital bed in the Central Zone was $1,101 (range $557-1,313).

By comparison, in a quality-improvement project on 750 inpatients with spinal cord injury in a large American hospital, Taylor et al. reported that patients with cervical-level injury had the highest mean wait times (8.28 days) for powered wheelchairs and the second highest was for manual rigid-frame wheelchairs (6.29 days). Other studies have found that the early mobilization of patients can lead to reductions in medical complications, lengths of stay and costs.

In summary, reductions in the Wheelchair Lead Time could speed patient mobilization (with benefits to the patient) and reduce the patient's hospital Length of Stay and the patient-related Cost of Hospitalization. However, at this time, these potential benefits remain speculative. The objectives for this Project are to test the hypotheses that there are positive correlations between Wheelchair Lead Time and both Length of Stay and the Cost of Hospitalization.

METHODS

Sample size Of the 119 patients available from the Pilot Study, the investigators plan to study all who meet the inclusion/exclusion criteria.

Database extraction The investigators will use the Medical Record Number and WheelEase order number to link, extract and deanonymize the data we need from the STAR (or Discharge Abstract), WheelEase, Capstone Pilot Study and Finance Department databases into an Excel file. The following data elements will be recorded in a common dataset: Medical Record Number, WheelEase order number, Date of birth, Sex, Diagnosis accounting for admission, Discharge destination, Order Origin, Order Date and time, Order Wheelchair type, Assembly Date and time, Delivery Date and time, and Hospital case cost.

Statistical analyses From the date of birth and order date, the investigators will calculate the age (in years) when the order was placed. From the dates for the Order, Assembly and Delivery events, the investigators will determine the days of the week corresponding to those dates. From the three events, three periods will be calculated: Wheelchair Assembly Time (from when ordered to assembled), Wheelchair Delivery Time (from when assembled to delivered) and Wheelchair Lead Time (from when ordered to delivered). All data will be reported descriptively. Where appropriate, the normality of the quantitative data will be assessed to guide the use of parametric vs nonparametric statistics. To test the hypotheses, the investigators will use Pearson or Spearman correlation coefficients. Secondarily, multivariate regression will be carried out with both Length of Stay and Cost of Hospitalization as dependent measures and age, sex, diagnosis, day of week that the order was placed (excluding weekends and holidays), site and wheelchair type as independent measures. The alpha level will be defined as 0.05. SAS statistical software will be used.

Economic analysis Hospital case cost includes all Nova Scotia Health direct, indirect and total costs (e.g., bed, lab, imaging, food, allied health, but excluding physician costs, operating-room supplies and days less than 24 hours) typically available up to the end of the prior fiscal year (March 31). Although the literature suggests that there should be positive patient outcomes resulting from any reductions in Wheelchair Lead Time, the investigators will not have data on such outcomes. Therefore, the economic analysis will be conducted from the perspective of the benefits to society. In any healthcare system with financial constraints, any system benefits must be weighed against their costs.

ELIGIBILITY:
Inclusion Criteria:

* to have been an inpatient in a Central Zone hospital site during the 11-weekday study period in late January 2023
* , to have had a WheelEase order placed during the 11-weekday study period in late January 2023
* to have had a Wheelchair Delivery Time recorded
* to have been subsequently discharged from a Central Zone hospital site.

Exclusion Criteria:

* if the WheelEase order was cancelled before delivery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in the Central Zone of Nova Scotia Health for whom a wheelchair was ordered using the WheelEase software.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Wheelchair Lead Time | Through initial study completion in 1 year
  Time from order placement to delivery to hospital site

SECONDARY OUTCOMES:
Length of stay | Through initial study completion in 1 year
  Duration of hospital admission
Case cost | Through initial study completion in 1 year
  Cost of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ronald L Kirby, MD, Principal Investigator — Dalhousie University
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No